CLINICAL TRIAL: NCT04690764
Title: Evaluation of the Effects of Preoperative Anxiety on Hemodynamics, Recovery and Drug Consumption in Patients Undergoing Total Intravenous Anesthesia (TIVA) for Neuromuscular Monitoring.
Brief Title: Evaluation of the Effects of Preoperative Anxiety in Patients Undergoing Total Intravenous Anesthesia (TIVA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Bülent Barış Güven, Anesthesiologist, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: 1423
Record Dates: First submitted 2020-12-27; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Preoperative Anxiety, Intraoperative Hemodynamics and Drug Consumption
Keywords: preoperative anxiety, total intravenous anesthesia,

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most patients have varying degrees of anxiety and fear before surgery. We believe that preopertive anxiety levels have an effect on intraoperative hemodynamics and recovery and affect intraoperative drug consumption. Inspired by this idea, we aimed to evaluate the effects of preoperative anxiety on hemodynamics, recovery, and drug consumption in patients undergoing total intravenous anesthesia (TIVA) due to neuromuscular monitoring.

DETAILED DESCRIPTION:
Introduction: Preoperative anxiety has been reported in 60-80% of the patients who will undergo surgery. Preoperative anxiety and fear may be due to the type of anesthesia, as well as to the patient's previous experiences, personality traits, concerns about surgical intervention, and postoperative pain. The anxiety levels of the patients can be affected by various factors such as their previous experiences, the way they come to the hospital, their gender, age, and the type of surgery they will undergo. The most widely used medical test for anxiety measurement is the State-Trait Anxiety Inventory (STAI) scale developed by Spielberg et al.

Objective: The primary aim of our study is to evaluate the effects of preoperative anxiety on intraoperative hemodynamics and recovery, and the secondary aim is to determine its effect on intraoperative drug consumption.

Hypothesis: Our hypothesis is that preoperative anxiety levels affect intraoperative hemodynamics and recovery and affect intraoperative drug consumption.

Materials and Methods: The study was planned prospectively, observationally. In the neurosurgery operating room of Sultan Abdülhamit Han Training and Research Hospital, patients whose operation is planned to be performed under neuromonitoring between 1 September 2019 and 1 February 2021 will receive a preoperative Spielberger State-Trait Anxiety Inventory (STAI) questionnaire and anxiety scores will be recorded. Afterward, routine anesthesia induction and follow-up will be performed for patients who are taken to the operating table. The preoperative anxiety score will be compared with the data recorded after the operation (hemodynamic data, total drug amount, recovery time).

Inclusion Criteria: Patients undergoing TIVA (Total Intravenous Anesthesia) due to Neuromuscular monitoring during neurosurgery operation, aged 18-70, who are literate, who do not have any psychiatric and neurological diseases, who are in ASA I and II class, Patients who do not drink alcohol regularly will be included in the study.

Exclusion Criteria: Patients who do not agree to participate in the study, patients who can not cooperate, patients using psychiatric drugs regularly and patients with chronic drug habits will be excluded from the study.

Study population: 80 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TIVA (Total Intravenous Anesthesia) due to Neuromuscular monitoring during neurosurgery operation, aged 18-70, who are literate, who do not have any psychiatric and neurological diseases, who are in ASA I and II class, Patients who do not drink alcohol regularly will be included in the study.

Exclusion Criteria:

* Patients who do not agree to participate in the study, patients who can not cooperate, patients using psychiatric drugs regularly and patients with chronic drug habits will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 Patients undergoing TIVA (Total Intravenous Anesthesia) due to Neuromuscular monitoring during neurosurgery operation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Spielberger State-Trait Anxiety Inventory (STAI) questionnaire and anxiety scores | Pre-surgery baseline to 1 week of postoperation
  STAI measures anxiety. The questionnaire asks the patients how they feel and allows them to respond on a frequency scale that ranges from 1(not at all) to 4(almost always/very much so). Scores range from 20-80 and the higher the score the greater the anxiety level.
Total intraoperative opioid consumption | During the neurological surgery
  The cumulative remifentanyl (microgram / kilogram) consumption after surgery will be recorded.
Total intraoperative propofol consumption | During the neurological surgery
  The cumulative propofol (miligram / kilogram) consumption after surgery will be recorded.

SECONDARY OUTCOMES:
Mean blood pressure change | within 5 minutes after surgical incision
  The maximal mean blood pressure within the first 5 minutes after surgical incision will be recorded.
  The mean blood pressure change from baseline will be calculated. The unit is mmHg.
Heart rate change | within 5 minutes after surgical incision
  The maximal heart rate within the first 5 minutes after surgical incision will be recorded.
  The heart rate change from baseline level will be calculated. The unit is beats per minute.
Lowest oxygen saturation | Time between neuromuscular blockade and 20 minutes after completion of endotracheal extubation
  Lowest oxygen saturation will be recorded and values under 95 percent will be considered low.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşın ERSOY, MD, Principal Investigator — Sultan Abdulhamidhan Training Hospital; bülent b güven, MD, Study Chair — Sultan Abdulhamidhan Training Hospital
Locations (1):
- Bülent Barış güven, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Maranets I, Kain ZN. Preoperative anxiety and intraoperative anesthetic requirements. Anesth Analg. 1999 Dec;89(6):1346-51. doi: 10.1097/00000539-199912000-00003. PMID 10589606
- [Result] Kim WS, Byeon GJ, Song BJ, Lee HJ. Availability of preoperative anxiety scale as a predictive factor for hemodynamic changes during induction of anesthesia. Korean J Anesthesiol. 2010 Apr;58(4):328-33. doi: 10.4097/kjae.2010.58.4.328. Epub 2010 Apr 28. PMID 20508787
- [Result] Ahmetovic-Djug J, Hasukic S, Djug H, Hasukic B, Jahic A. Impact of Preoperative Anxiety in Patients on Hemodynamic Changes and a Dose of Anesthetic During Induction of Anesthesia. Med Arch. 2017 Oct;71(5):330-333. doi: 10.5455/medarh.2017.71.330-333. PMID 29284900